CLINICAL TRIAL: NCT05844228
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of VIR-2218 in Adult Participants With Renal Impairment
Brief Title: A Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics and Safety of VIR-2218
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-2218-V108
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Up to 8 moderate Renal Impairment (RI) participants and 8 matched healthy participants (Experimental)
  Interventions: Drug: VIR-2218
- Cohort 2: Up to 8 severe Renal Impairment (RI) participants and 6 matched healthy participants (Experimental)
  Interventions: Drug: VIR-2218

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
  Other Names: Elebsiran

SUMMARY:
The rationale of this study is to evaluate the impact of renal function on the PK, safety, and tolerability of VIR-2218 in participants with normal renal function and participants with varying degrees of renal dysfunction who are otherwise medically stable

DETAILED DESCRIPTION:
Participants may be enrolled in Cohorts 1 and 2 in a non-randomized way.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Participants must have stable renal function as defined by less than 20% change in estimated glomerular filtration rate (eGFR) between the first and second screening sample with the first screening visit occurring within 28 days prior to dosing on Day 1 and the second screening visit occurring no more than 14 days apart, but at least 72 hours apart from the first.
* Body mass index (BMI) within the range 18.5 to 40.0 kg/m^2 at screening.
* Female and Male participants must consent to follow contraception requirements
* Capability of giving signed informed consent form

Inclusion Criteria: Additional Criteria Specific to Healthy Participants:

* Must be in the opinion of the investigator, be in good health based upon medical history, vital signs, physical examination, and screening laboratory evaluations
* Must have normal renal function as defined by eGFR ≥ 90 mL/min/1.73m^2 based on the Modification of Diet in Renal Disease (MDRD) equation determined from the mean of two measurements of serum creatinine at screening.

Inclusion Criteria: Additional Criteria Specific to Participants with Renal Impairment

* Participants must, in the opinion of the investigator, be sufficiently healthy for study participation based on medical history, physical examination, vital signs, and screening laboratory evaluations
* Participants with RI must have chronic moderate or severe RI and be clinically stable per investigator assessment for at least 3 months prior to screening
* Moderate RI as defined by eGFR level 30-59 mL/min/1.73m^2 based on the MDRD equation, or
* Severe RI as defined by eGFR level 15-29mL/min/1.73m^2 based on the MDRD equation

Exclusion Criteria: Criteria for All Participants

* Any clinically significant medical condition or psychiatric condition that may interfere with study intervention
* Participants with uncontrolled hypertension, asthma, and/or diabetes (Type I or II).
* Participants with diabetes
* Participants with any active malignancy
* Participants with vasculitis or conditions associated with vasculitis.
* Participants who have undergone major surgery within 12 months of screening
* Participants with unstable cardiac functions, abnormality, or clinically significant heart failure
* Participants with infection of HIV, HAV, HBV, HCV, HDV, or HEV
* Participants with signs of active infection
* History of bone marrow or solid organ transplantation
* Participants with end-stage renal disease or nephrotic syndrome as defined by: participants requiring hemodialysis or peritoneal dialysis, participants who have undergone or are listed for transplant, or participants who have chronic kidney disease with nephrotic syndrome
* Participants with active nephritis
* Participants with clinically significant liver disease
* History of drug or alcohol abuse
* Unwillingness or inability to follow procedures outlined in protocol

Exclusion Criteria: Additional Criteria Specific to Healthy Participants

* Use of any prescription medications or over-the-counter medications (with the exception of vitamins and/or hormonal contraceptive medications) including herbal products within 30 days prior to D1 of study participation

Exclusion Criteria: Additional Criteria Specific to Participants with Renal Impairment

* Not on stable dose and regimen of any medication(s) (prescription or over-the-counter) that the participants is taking regularly (eg, medications for chronic conditions such as hypertension, high cholesterol, or depression must not be changed in dose or type for at least 2 weeks prior to study drug administration). Use of other prescription medications or over-the-counter medications that are not for chronic conditions (with the exception of vitamins and/or hormonal contraceptive medications) including herbal products within 30 days prior to D1 of study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days
Area Under The Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUClast) of VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days
Fraction excreted in urine in percentage for VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days
Amount excreted in urine for VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days
Renal clearance for VIR-2218 and its metabolite AS(N-1)3'VIR-2218 | 5 days

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Inland Empire Clinical Trials, Rialto, California
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida